CLINICAL TRIAL: NCT04052048
Title: A Multi-center, Prospective Active Surveillance Registry Trial Assessing the Performance of a Non-invasive Immunogenomic Blood Test for Indolent Prostate Cancer Disease Management.
Brief Title: Active Surveillance SNEP Assay Registry Trial for Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Immunis.AI (Industry)
Responsible Party: Sponsor
Other Study IDs: ONC-AS-2019
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer Aggressiveness
MeSH Terms: conditions — Prostate Cancer, Hereditary, 7

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Three tubes of blood:
  Two 8ml CPT One 4ml SST
  Prostate Biopsy slides
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Subtraction Normalized Expression of Phagocytes Blood Test — Non-invasive blood based immunogenomic assay that targets RNA sequencing to identify disease and disease aggressiveness

SUMMARY:
A multi-center, prospective active surveillance registry trial assessing the performance of a non-invasive blood test for indolent prostate cancer disease management.

DETAILED DESCRIPTION:
The analysis population is defined as all the set of de-identified patient results received from the practices who met the inclusion / exclusion criteria. A target recruitment of 2000 subjects with an expected loss of 20% (400 subjects) and an overall event rate of 30% (480 subjects of 1600) will result in 480 cases and 1120 controls, where cases are defined as those patients with NCCN unfavorable intermediate risk or worse disease. With a significance level alpha of 0.05, the number of cases above will result in a statistical power (1-ß=0.2) of at least 80% to show a significant increase in performance of the full assay over clinical variables alone, assuming that performance characteristics are similar to those observed in a retrospective, independent training cohort and that the patients in the SAFELY cohort resemble this same training population.

ELIGIBILITY:
Inclusion Criteria

* Men between 40-80 of age with at least a 10-year life expectancy
* All active surveillance protocols are accepted
* No PSA limits

Category 1:

* Patient is currently on active surveillance with only ONE previous low grade prostate biopsy.
* Patient must already be scheduled for their 1st annual biopsy under their active surveillance protocol within 90 days of enrollment date.

Category 2:

• Patient is recently diagnosed with low grade prostate cancer but has decided against active surveillance and is scheduled for radical prostatectomy within 90 days of enrollment date.

Exclusion Criteria:

Men on watchful waiting i.e. those with less than 10-year life expectancy with no intent for curative therapy

* Men with symptoms or rising PSA who have not been proven to have cancer by tissue biopsy i.e. men with only negative prostate biopsies.
* Patients with a history of a different cancer (except basal cell carcinoma)

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer who are on or are candidates for Active surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Collect performance results on assay's ability to identify occult aggressive disease in active surveillance population. | 1 year
  Collect information from repeat biopsy including any increase in gleason grade, increase in number of cores positive, and increase in % cross sectional surface area involved by tumor from the repeat biopsy.

SECONDARY OUTCOMES:
Validate immunogenomic assay's ability to serve as an ongoing, non-invasive tool to monitor patient risk for disease progression as detected by repeat biopsy. | 10 years
  On an annual basis, collect follow-up frequency data for each patient including optional repeat blood testing, repeat biopsy data, disease management decisions, and disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Urology, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmer C, Diehn M, Alizadeh AA, Brown PO. Cell-type specific gene expression profiles of leukocytes in human peripheral blood. BMC Genomics. 2006 May 16;7:115. doi: 10.1186/1471-2164-7-115. PMID 16704732
- [Background] Schmidl C, Renner K, Peter K, Eder R, Lassmann T, Balwierz PJ, Itoh M, Nagao-Sato S, Kawaji H, Carninci P, Suzuki H, Hayashizaki Y, Andreesen R, Hume DA, Hoffmann P, Forrest AR, Kreutz MP, Edinger M, Rehli M; FANTOM consortium. Transcription and enhancer profiling in human monocyte subsets. Blood. 2014 Apr 24;123(17):e90-9. doi: 10.1182/blood-2013-02-484188. Epub 2014 Mar 26. PMID 24671955
- [Background] Hashimoto S, Nagai S, Sese J, Suzuki T, Obata A, Sato T, Toyoda N, Dong HY, Kurachi M, Nagahata T, Shizuno K, Morishita S, Matsushima K. Gene expression profile in human leukocytes. Blood. 2003 May 1;101(9):3509-13. doi: 10.1182/blood-2002-06-1866. Epub 2003 Jan 9. PMID 12522010
- [Background] Dale DC, Boxer L, Liles WC. The phagocytes: neutrophils and monocytes. Blood. 2008 Aug 15;112(4):935-45. doi: 10.1182/blood-2007-12-077917. PMID 18684880
- [Background] Gutknecht MF, Bouton AH. Functional significance of mononuclear phagocyte populations generated through adult hematopoiesis. J Leukoc Biol. 2014 Dec;96(6):969-80. doi: 10.1189/jlb.1RI0414-195R. Epub 2014 Sep 15. PMID 25225678
- [Background] Chow A, Brown BD, Merad M. Studying the mononuclear phagocyte system in the molecular age. Nat Rev Immunol. 2011 Oct 25;11(11):788-98. doi: 10.1038/nri3087. PMID 22025056
- [Background] Epstein JI. An update of the Gleason grading system. J Urol. 2010 Feb;183(2):433-40. doi: 10.1016/j.juro.2009.10.046. Epub 2009 Dec 14. PMID 20006878
- [Background] Grignon DJ. Prostate cancer reporting and staging: needle biopsy and radical prostatectomy specimens. Mod Pathol. 2018 Jan;31(S1):S96-109. doi: 10.1038/modpathol.2017.167. PMID 29297497
- [Background] Boutros PC, Fraser M, Harding NJ, de Borja R, Trudel D, Lalonde E, Meng A, Hennings-Yeomans PH, McPherson A, Sabelnykova VY, Zia A, Fox NS, Livingstone J, Shiah YJ, Wang J, Beck TA, Have CL, Chong T, Sam M, Johns J, Timms L, Buchner N, Wong A, Watson JD, Simmons TT, P'ng C, Zafarana G, Nguyen F, Luo X, Chu KC, Prokopec SD, Sykes J, Dal Pra A, Berlin A, Brown A, Chan-Seng-Yue MA, Yousif F, Denroche RE, Chong LC, Chen GM, Jung E, Fung C, Starmans MH, Chen H, Govind SK, Hawley J, D'Costa A, Pintilie M, Waggott D, Hach F, Lambin P, Muthuswamy LB, Cooper C, Eeles R, Neal D, Tetu B, Sahinalp C, Stein LD, Fleshner N, Shah SP, Collins CC, Hudson TJ, McPherson JD, van der Kwast T, Bristow RG. Spatial genomic heterogeneity within localized, multifocal prostate cancer. Nat Genet. 2015 Jul;47(7):736-45. doi: 10.1038/ng.3315. Epub 2015 May 25. PMID 26005866
- [Background] Womble PR, Montie JE, Ye Z, Linsell SM, Lane BR, Miller DC; Michigan Urological Surgery Improvement Collaborative. Contemporary use of initial active surveillance among men in Michigan with low-risk prostate cancer. Eur Urol. 2015 Jan;67(1):44-50. doi: 10.1016/j.eururo.2014.08.024. Epub 2014 Aug 24. PMID 25159890
- [Background] Cher ML, Dhir A, Auffenberg GB, Linsell S, Gao Y, Rosenberg B, Jafri SM, Klotz L, Miller DC, Ghani KR, Bernstein SJ, Montie JE, Lane BR; Michigan Urological Surgery Improvement Collaborative. Appropriateness Criteria for Active Surveillance of Prostate Cancer. J Urol. 2017 Jan;197(1):67-74. doi: 10.1016/j.juro.2016.07.005. Epub 2016 Jul 14. PMID 27422298